CLINICAL TRIAL: NCT05691335
Title: Analysis of the Outcomes of Three Different Cross-linking Protocols for Treatment of Pediatric Keratoconus
Brief Title: Three Different Cross-linking Protocols for Treatment of Pediatric Keratoconus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Prof. Mohammed Iqbal, Professor, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10-4/2018
Record Dates: First submitted 2023-01-07; First posted 2023-01-20 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Corneal Ectasia
MeSH Terms: interventions — Corneal Cross-Linking

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard CXL (Other): Patients treated according to Dresden Protocol with epithelium-off CXL.
  Interventions: Procedure: Standard CXL
- Accelerated CXL (Experimental): Patients treated according to accelerated Protocol with epithelium-off CXL.
  Interventions: Procedure: Accelerated CXL
- Transepithelial CXL (Experimental): Patients treated according to transepithelial Protocol with epithelium-on CXL.
  Interventions: Procedure: Transepithelial CXL

INTERVENTIONS:
Procedure: Standard CXL — Epithelium-off CXL performed by removal of corneal epithelium, instillation of riboflavin onto the cornea followed by UVA corneal irradiation for 30 minutes.
  Arms: Standard CXL
Procedure: Accelerated CXL — Epithelium-off CXL performed by removal of corneal epithelium, instillation of riboflavin onto the cornea followed by UVA corneal irradiation for 5 minutes.
  Arms: Accelerated CXL
Procedure: Transepithelial CXL — Epithelium-on CXL performed by instillation of riboflavin onto the cornea followed by UVA corneal irradiation for 5 minutes.
  Arms: Transepithelial CXL

SUMMARY:
comparison between standard cross-linking protocol and accelerated and transepithelial cross-linking

DETAILED DESCRIPTION:
comparison between standard cross-linking protocol and accelerated and transepithelial cross-linking for treatment of documented pediatric keratoconus progression. The study patients are divided into 3 groups. Group A patient treated with standard cross-linking. Group B patients treated with accelerated cross-linking. Group C patients treated with transepithelial cross-linking.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patient less than 18 years old
* keratoconus stage I-III ABCD keratoconus grading system

Exclusion Criteria:

* age more than 18 years
* previous eye surgery
* current eye infection or pathology

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 97 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-05 (Actual)

PRIMARY OUTCOMES:
Uncorrected distance visual acuity | 36 months
  measured in logarithm of minimal angle of resolution (logMAR)
Corrected distance visual acuity | 36 months
  measured in logarithm of minimal angle of resolution (logMAR)
Sphere | 36 months
  measured in diopters (D)
Cylinder | 36 months
  measured in diopters (D)
Keratometry (Kmax) | 36 months
  measured in diopters (D)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Iqbal, MD, PhD, Principal Investigator — Sohag University
Locations (1):
- Faculty of medicine, Sohag, Egypt